CLINICAL TRIAL: NCT07065305
Title: Clinical Performance and Remineralization Potential of Self- Assembling Peptide P11-4 Containing Fluoride Versus Er, Cr: YSGG Laser Treatment and Micro Tensile Bond Strength of Giomer Restoration in Carious Lesions
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Fatheya Mansour Elshinawy, Assistant lecturer of Restorative Dentistry, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPDEN-103-1-S
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Remineralization Potential; Dentin Caries
Keywords: Er, Cr: YSGG Laser; Caries-Affected Dentin; Remineralization Potential; Self-Assembling Peptide P11-4 Containing Fluoride
MeSH Terms: interventions — Fluorides; Bisphenol A-Glycidyl Methacrylate; triethylene glycol dimethacrylate

STUDY DESIGN:
Intervention Model Description: * Group 1 no pretreatment will received.
  * Group 2 will receive Curodont Repair (P11-4 plus fluoride).
Who Masked: Participant
Masking Description: * Eligible patients will be randomly assigned to the intervention or control group using computer-generated random numbers.
  * Allocation concealment will be ensured using sealed opaque envelopes.
  * Clinical evaluators assessing outcomes will be blinded to the group allocation to reduce bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curodont Repair Fluoride Plus (P11-4 + fluoride) (Experimental): • In the Intervention group the Curodont Repair (P11-4 + fluoride) will be applied according to the manufacturer's instructions: The paste is gently applied to the dentin surface and left undisturbed for 5 minutes to allow self-assembly and infiltration and excess material will be removed with a gentle air spray
  Interventions: Drug: Curodont Repair Fluoride Plus (Self-assembling peptide remineralization agent)P11-4 peptide, fluoride, mild acidic buffer (pH ~4.5) , Credentis AG, Switzerland; Drug: Beautifil II LS
- Beautifil II LS (Placebo Comparator): No pretreatment; proceed directly to bonding. Then the surface will dry with absorbent paper. A layer of the adhesive system (BeautiBond extrem, Shofu Inc., Kyoto, Japan) will be actively applied for 20 seconds using a micro brush. Then, the adhesive will light-cure for 10 seconds with Radii-cal LED light curing device (1200 mW/cm2) (SDI, Bayswater, Australia) (2
  Interventions: Drug: Curodont Repair Fluoride Plus (Self-assembling peptide remineralization agent)P11-4 peptide, fluoride, mild acidic buffer (pH ~4.5) , Credentis AG, Switzerland; Drug: Beautifil II LS

INTERVENTIONS:
Drug: Curodont Repair Fluoride Plus (Self-assembling peptide remineralization agent)P11-4 peptide, fluoride, mild acidic buffer (pH ~4.5) , Credentis AG, Switzerland — Pretreatment with Curodont Repair Fluoride Plus (P11-4 + fluoride)
Drug: Beautifil II LS — Application of Giomer restorative material following standard adhesive procedures without pretreatment.
  Other Names: S-PRG (Surface Pre-Reacted Glass-ionomer) filler, Bis-GMA, TEGDMA, glass fillers , Shofu Inc., Kyoto, Japan; Giomer-based restorative composite

SUMMARY:
This study will be performed in two parts, in vivo and in vitro to assess the effect of the remineralization potential of self-assembling peptide P11-4 containing Fluoride on caries-affected dentin compared to untreated caries-affected dentin and the influence of Er, Cr: YSGG Laser treatment.

DETAILED DESCRIPTION:
The present study will be performed to evaluate the remineralization potential of the self-assembling peptide P11-4 combined with fluoride treatment applied over demineralized dentin in occlusal carious molars.

* Research objectives: To assess the effect of the two treatment modalities to enhance remineralization of demineralized dentin and clinical performance of restorations.
* Research question: Will pretreatment of caries affected dentin using self-assembling peptide P11-4 containing fluoride compared to untreated caries-affected dentin will enhance the remineralization and clinical performance of composite restorations In Vitro Study

  1- The present study will be performed to evaluate the remineralization potential of the self-assembling peptide P11-4 combined with fluoride and its effect on bond strength and analyze morphological changes over demineralized dentin in occlusal carious molars using Scanning Electron Microscopy (SEM).
* Research Objectives: To evaluate the effect of Curodont Repair Fluoride Plus and Er,Cr:YSGG laser pretreatment on the bond strength of composite resin to superficial and deep dentin.
* Research question: Will pretreatment of caries affected dentin using self-assembling peptide P11-4 containing fluoride compared to untreated caries-affected dentin will enhance bond strength?

ELIGIBILITY:
Inclusion Criteria:

* o Patients aged (20 - 40) years.

  * Presence of at least one posterior permanent molar with an occlusal carious lesion classified as ICDAS code 3 or 4 requiring operative treatment.
  * Good general and oral health.
  * Willingness to participate and provide informed consent.

Exclusion Criteria:

* o Patients with systemic conditions affecting oral health or healing.

  * Teeth with pulp involvement or periapical pathology.
  * Allergy to study materials.
  * Poor oral hygiene or periodontal disease in the target tooth region.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Marginal integrity of restorations | 6 months and 12 months
  Assessed using mirror and probe according to Modified USPHS Criteria
Clinical longevity of restorations | 6 and 12 months
  Assessed by restoration retention using mirror and probe
Overall clinical performance of restorations | 6 and 12 months
  Evaluated using Modified USPHS Criteria

SECONDARY OUTCOMES:
Postoperative hypersensitivity | 6 and 12 months
  Evaluated using cold spray test
Marginal discoloration | 6 and 12 months
  Assessed using digital photographic method
Recurrent caries | 6 and 12 months
  Detected using digital photographic method
Surface roughness | 6 and 12 months
  Evaluated using digital photographic method
Surface luster | 6 and 12 months
  Assessed using digital photographic method